CLINICAL TRIAL: NCT00288600
Title: Phase 4 Study of Use of High-dose Intravenous Immune Globulin for Prevent Hyperbilirubinemia Due Rh Hemolytic Disease in Newborns Infants
Brief Title: Efficacy of High-dose Intravenous Immunoglobulin Therapy for Hyperbilirubinemia Due Rh Hemolytic Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Instituto Fernandes Figueira (Other Government)
Responsible Party: Principal Investigator, Maria Elisabeth Lopes Moreira, MD, PhD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ivig01
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Hyperbilirubinemia; Erythroblastosis, Fetal
Keywords: Immunoglobulins, Intravenous; Hyperbilirubinemia; Erythroblastosis, Fetal; Exchange Transfusion, Whole Blood
MeSH Terms: conditions — Hyperbilirubinemia; Erythroblastosis, Fetal | interventions — Immunoglobulins, Intravenous; Immunoglobulins; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Intravenous Immunoglobulin
  Interventions: Drug: Intravenous Immunoglobulin
- CONTROL GROUP (Placebo Comparator): Normal Saline solution
  Interventions: Drug: Normal saline solution

INTERVENTIONS:
Drug: Intravenous Immunoglobulin — Intravenous Immunoglobulin
  Other Names: Immunoglobulin
  Arms: Experimental group
Drug: Normal saline solution — Normal saline solution 10 ml/Kg
  Other Names: saline solution
  Arms: CONTROL GROUP

SUMMARY:
The use of intravenous immunoglobulin G (IVIG) therapy has been reported in hyperbilirubinemia of Rh hemolytic disease but we don't have enough evidences for it. Human Immunoglobulin is considered an alternative to delay the hemolytic process and consequently reduce the number of exchange transfusions and transfusions of red cells concentrate, thus diminishing the risk of transmitting transfusional therapies-related diseases. OBJECTIVE: To determine the effect of IVIG in decreasing the incidence and severity of neonatal immune hemolytic jaundice due to Rh hemolytic disease reducing the need for exchange transfusion as a primary goal in these babies. METHODS: This will be a randomized, double blind, clinical trial involving all newborns with risk of significant hyperbilirubinemia due to direct Coombs-positive Rh hemolytic disease. The primary goal will be need for exchange transfusion and others are: incidence of late anemia, kernicterus and deafness Babies were randomly assigned into two groups: group 1 (study group) received phototherapy plus IVIG (500 mg/kg); and group 2 (control group) received phototherapy and normal saline solution (10 ml/Kg) in the first 6 hours of life. Exchange transfusion was carried out in any group if at any time the bilirubin level reached 340 micromol/l (20 mg/dl) or more, or rose by 8.5 micromol/l per h (0.5 mg/dl per h). Adverse effects will be related in two groups. Parents informed consent will be asked in pre-natal time.

DETAILED DESCRIPTION:
The Hemolytic Anemia due to Rh alloimmunization is characterized by the hemolysis of Rh (D) fetal red cells caused by the action of anti Rh (D) maternal antibodies in the fetal circulation.

The perinatal hemolytic disease due to Rh alloimmunization is almost extinct all over the world. The administration of Specific Human Immunoglobulin prevents the sensitization process and when introduced in the perinatal care of pregnant women, it reduces the incidence of cases of Rh alloimmunization.

Unfortunately Brazil does not have effective policies geared to reducing the perinatal hemolytic disease and its consequences and thus the incidence of this condition continues to be high.

The conventional treatment includes phototherapy and exchange transfusion. The advantages of the exchange transfusion in the Rh hemolytic disease are well defined but its risks remain high and the mortality rates related to the procedure range around 2% and the morbimortality (thrombocytopenia, thrombosis of the portal vein, necrotizing enterocolitis, metabolic disorders and infection) reach 12%. The procedure requires the availability of compatible blood, a team with appropriate training in the procedure and a neonatal ICU infrastructure prepared to prevent the admission of newborns whose mothers did not go through prophylaxis.

The use of immunoglobulin associated to phototherapy may reduce the need for exchange transfusion, thus allowing for more sensitized newborns to receive treatment and therefore avoiding neurological damages associated with the hemolytic disease.

If the high incidence of the disease, the difficulties and the risks involved in an exchange transfusion, the difficulties in obtaining Rh negative blood are taken into consideration, it becomes clear that it is important conducting studies to prove the effectiveness of the immunoglobulin in such cases.

General Objective To determine the effect of IVIG in decreasing the incidence and severity of neonatal immune hemolytic jaundice due to Rh hemolytic disease reducing the need for exchange transfusion as a primary goal in these babies.

Specific Objectives

1. To asses if the administration of immunoglobulin in newborns with hyperbilirubinemia caused by alloimmunization Rh(D) hemolytic anemia:

   1. Reduces the need for phototherapy
   2. Reduces the length of the phototherapy treatment
   3. Reduces the need or number of exchange transfusion
   4. Reduces the time of hospitalization
2. To evaluate the risk for those patients that received immunoglobulin and the side effects during its administration.
3. To evaluate the incidence of late anemia and the sequelae of hyperbilirubinemia (deafness, development retardation, cholestasis and kernicterus) during the first year of life.
4. To evaluate the Ig-G subclasses and the presence of anti-HLA antibodies of paternal blood cells in the groups of newborns studied and their relation with the clinical response to immunoglobulin.

Methodology This will be a randomized and double-blind clinical trial essay . The mothers will be approached during the prenatal treatment, after being diagnosed as carriers of hemolytic disease due to Rh alloimmunization. The research will be presented and the mother/family will be invited to participate in the study. The informed consent term will be presented to the mother/family and they will be allowed some time to decide. If they are accepted in the study they will receive a questionnaire on the issues related to the possible reasons of sensitization.

After obtaining the free and informed consent from the parents, the sensitized newborns will be randomized in 2 groups, in a 1:1 proportion. The study group will receive Human Immunoglobulin (Immunoglobulin® - 50mg/ml) with a dose of 500mg/kg, equivalent to 10ml/kg during the initial 6hours of life, through intravenous infusion for 2 hours; the control group will receive the same volume in saline solution at 0.09%.

All newborns included in the study will be granted with conventional supplementary treatment that includes the indication of exchange transfusion and of phototherapy, according to specific criteria recommended by the American Academy of Pediatrics in 2004. The criteria apply equally to both groups. The study will be monitored individually and it will be allowed to be interrupted it if any important side effect occurs such as anaphylactic reaction or if the results of a given group are significantly better than those of the other before the inclusion of new subjects in the research, according to the size of the sample or in case the drug does not yield the desired beneficial effects.

An independent neonatologist, previously chosen, will check the undesirable side effects and will partially monitor the results of the study. The report on undesirable effects will be conducted for each case; two intermediate evaluations on the results of the research are to be conducted. The Committee on Ethics on Research will be informed of every non-expected or undesired effect related to the medication under study or of the need to interrupt the research.

Sample Size :

The calculated size of the sample, considering a reduction of 30% on the indication of exchange transfusion, with a statistical significance of 95% and test power of 80% was 90 newborns. An investigator will approach all pregnant women and/or parent/responsible for the babies potentially eligible for the study and he will deliver them a consent term.

Randomization and blinding The randomization will be performed by drawing blocks of different sizes. In order to avoid that the health professionals in the nursery know which product is being infused into the newborns (Immunoglobulin or Saline Solution 0.9%) the syringes with the required volumes will be prepared in the pharmacy and wrapped in aluminum foil. The color of the products is similar. The newborns will be monitored and clinically followed-up before, during and after the two groups equally receive the infusion. All clinical changes such as cardiac and respiratory frequency and hemoglobin saturation will be recorded before and after the infusion in the two groups. All newborns, before and after the procedure, will be submitted to Glucose dosages by screening method (Blood sugar test).

Complementary treatment

The complementary treatment will be administered and secured to all newborns admitted into the study and will follow the protocols below:

Indication for exchange transfusion

The babies to whom an exchange transfusion at birth would be indicated will be excluded from the study. The indications for exchange transfusion at birth are:

* Bilirubin on the umbilical cord superior or equal to 4 mg%
* Fetal hydrops or congestive heart failure due to serious anemia.

The exchange transfusion will be indicated to the following newborns after birth, according to the existing literature and presenting the following features:

* Bilirubin level is rising over 0.5mg/dl per hour despite phototherapy or
* Hyperbilirubinemia, according to APP directives.

Indication of Phototherapy

All newborns will receive phototherapy beginning in the first 6 hours of life The procedure adopted will be the triple phototherapy placed 50cms away from the newborns; the irradiance of the device will be measured every day.

Indication for blood transfusion:

The newborns that present the conditions mentioned below will be indicated to receive reed blood transfusion at the volume of 15ml/kg, according to criteria below:

1. Hematocrit level under 25% with positive direct or indirect Coombs Hematocrit level under 21%, with negative direct and indirect Coombs
2. Reticulocytes - less than 1%
3. Hematocrit level under 30% accompanied by clinical signs of severe anemic. Auditory Evoked Potential All newborns involved in the study will undergo a non-invasive hearing test, at the occasion of hospital discharge or at the first time they go to the ambulatory for follow-up. The application of the hearing evoked potential is indicated to all isoimmunized newborns and is routinely performed at the local where the study is taking place.

Follow-up after hospital discharge All newborns will be followed-up at the Follow-Up Ambulatory until the first year of life, during which the laboratorial follow-up will be conducted (Hematocrit/Coombs) as well as the complete physical and neurological examination. The Bayley method will be used for neurological evaluation, to be performed by a trained professional at the end of the first year of life. Every fact related to the clinical evolution during the first year of life will be recorded: the presence of cholestasis, nutritional situation (evaluation) through z-score at the time of hospital discharge, by the 6th month and at the end of the first year, regarding weight, height and head perimeter, using NCHS as standard; hospital admittance for blood transfusion or other treatments, presence of infection that might be related to the use of blood derivates (hepatitis B and C , cytomegalovirus).

Laboratorial Tests The laboratorial exams will be performed based on maternal samples, drawn during the pre-natal period and on samples of the newborn, drawn at birth (blood of the umbilical cord) and through heel puncture and withdrawal of 2 capillary tubes. These capillaries will be centrifuged and the total bilirubin will be measured by the Bilirubin Meter B105, ERMA INC.). The technicians to perform the exams will not be aware of the allocated group of the patient under examination.

1. Determination of ABO blood groups of the mother- direct and reversal proof- a technique in the vial with BIOTEST reagents.
2. Determination of the ABO blood group of the newborn -
3. Determination of maternal and fetal Rho ( D) factor - Technique in vial using the anti-D monoclonal saline solution and BIOTEST Rh control saline solution.
4. Research for irregular antibodies P.A I - in the phase of immediate reading, proteic phase at 37º - technique in the vial with BIOTEST reagents and sensitized red cell-test ( Coombs control) by BIOTEST
5. Identification of Irregular Antibodies - technique performed with reagents in the albuminous Coombs vial and a Panel of phenotyped red cells and sensitized red cells ( Combs Control) by BIOTEST
6. Dosage of irregular antibodies in the maternal serum with phenotyped red cells of the newborn
7. Research for anti-A and anti-B IgG in the blood serum of the Rh negative alloimmunized, blood type "O" positive mother.
8. Direct test of human immunoglobulin (Direct Coombs) in samples of the NB - technique performed in a vial with BIOTEST reagents.
9. Classification of IgG subclasses - immunoenzymatic test (ELISA)
10. Research for anti-HLA antibodies against paternal blood cells.

Data analysis:

The data will be stored in the attached worksheet and analyzed using statistical methods to compare the results of laboratorial exams and the presence or absence of exchange transfusion during hospital stay among those children who were given intravenous immunoglobulin and those that were not. These tests will take into consideration that the sample has been randomized in blocks. The observations will also be conducted by stratifying both groups, as follows: premature babies, non-premature babies, babies that underwent intra-uterus transfusion and those that did not. The data will be examined by the statistical program SPSS 13.0, using the appropriate tests for quantitative and binary variables.

ELIGIBILITY:
Inclusion Criteria:

* All newborns with a gestational age equal or higher than 32 weeks, with a Rh (D) positive blood type, children of sensitized Rh (D) negative mothers, regardless if they were submitted or not to an intra-uterus transfusion.

Exclusion Criteria:

* Newborns in serious condition, hydropic, hemodynamically instable or with indication for exchange transfusion at birth. The indications for exchange transfusion at birth are: presence of bilirubin in the umbilical cord higher or equal to 4mg%; hydrops, cardiac insufficiency secondary to severe anemia.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria EL Moreira, MD, Principal Investigator — Oswaldo Cruz Foundation
Locations (1):
- Maria Elisabeth L Moreira, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Santos MC, Sa C, Gomes SC Jr, Camacho LA, Moreira ME. The efficacy of the use of intravenous human immunoglobulin in Brazilian newborns with rhesus hemolytic disease: a randomized double-blind trial. Transfusion. 2013 Apr;53(4):777-82. doi: 10.1111/j.1537-2995.2012.03827.x. Epub 2012 Aug 6. PMID 22882285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessed for eligibility 125
  Excluded (n= 33) Not meeting inclusion criteria (n= 26) Declined to participate (n= 4) Other reasons (n= 3)
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 46 | 46
Completed | 46 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group - Immunoglobulin: Intravenous Immunoglobulin and Phototherapy
  Intravenous Immunoglobulin: Intravenous Immunoglobulin
- Control Group- Normal Saline: Normal Saline solution and Phototherapy
  Normal saline solution: Normal saline solution 10 ml/Kg
- Total: Total of all reporting groups
Arm/Group | Experimental Group - Immunoglobulin | Control Group- Normal Saline | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Median (Full Range); unit: hours of life] | 3 [1 to 4.5] | 3 [1 to 4.2] | 3 [1 to 4.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 26 | 23 | 49
Region of Enrollment [Number; unit: participants]
  Brazil | 46 | 46 | 92
maternal age [Mean (Standard Deviation); unit: years] | 30.6 (6.0) | 30.0 (6.2) | 30.2 (6.2)
TSB at birth [Mean (Standard Deviation); unit: mg/dl] | 2.42 (1.29) | 2.87 (1.49) | 2.64 (1.36)

OUTCOME MEASURES:

1. Primary Outcome: Need of Exchange Transfusion
Description: NEED OF EXCHANGE TRANSFUSION FOLLOWING GUIDELINES
Time Frame: 10 DAYS OF LIFE
Population: NUMBER
Measure: Number; unit: participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 46 | 46
participants | 6 | 7
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Need of Exchange transfusion following the AAP criteria; Test type: Superiority or Other; p = 0.765, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

LIMITATIONS AND CAVEATS:
We calculated the sample size using a expected rate of 30% reduction in exchange using incidence of exchange transfusion at our department and data from a meta-analysis (relative risk, 0.21; 95% CI 0.10-0.45).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No